CLINICAL TRIAL: NCT01404533
Title: The Influence of Iron Interventions on Formation of Non-transferrin-bound Iron (NTBI) in Women
Brief Title: Iron Interventions and Non-transferrin-bound Iron (NTBI) in Women
Acronym: NTBIwomen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NTBI women
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Iron Deficiency
Keywords: NTBI; Iron; Absorption
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Iron supplement without food (Experimental)
  Interventions: Dietary Supplement: Ferrous sulfate
- Iron supplement with food (Experimental)
  Interventions: Dietary Supplement: Ferrous sulfate
- Iron fortificant with food (Experimental)
  Interventions: Dietary Supplement: Ferrous sulfate

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate — 60 mg Ferrous sulfate
  Arms: Iron supplement without food
Dietary Supplement: Ferrous sulfate — 60 mg ferrous sulfate
  Arms: Iron supplement with food
Dietary Supplement: Ferrous sulfate — 6 mg ferrous sulfate
  Arms: Iron fortificant with food

SUMMARY:
The overall goal of this research is to develop safe and effective iron interventions that can be administered without production of plasma non-transferrin-bound iron (NTBI: iron in the systemic circulation not bound to the iron-transport protein transferrin). The appearance of plasma non-transferrin-bound iron has been reported in uninfected adult volunteers after oral administration of iron supplements in doses similar to those used in the Pemba trial. This research project will (i) confirm the appearance of plasma non-transferrin-bound iron after administration of an iron supplement like that in the Pemba trial (~1 mg Fe/kg body weight, without food), and then determine the effects on production of plasma non-transferrin-bound iron and on iron absorption measured with stable isotopes (ii) of giving the supplemental iron (~1 mg Fe/kg) with the standard rice meal, and (iii) of giving a lower dose of iron (~0.1 mg Fe/kg) - like that used in home fortification - with the standard rice meal.

ELIGIBILITY:
Inclusion Criteria:

* non pregnant
* non lactating
* apparently healthy women

Exclusion Criteria:

* chronic disease
* pregnancy
* lactation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Formation of NTBI following oral iron administration | 6 time points within 8 hours

SECONDARY OUTCOMES:
Serum iron isotope appearance curves | 6 time points within 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hurrell, PhD, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Brittenham GM, Andersson M, Egli I, Foman JT, Zeder C, Westerman ME, Hurrell RF. Circulating non-transferrin-bound iron after oral administration of supplemental and fortification doses of iron to healthy women: a randomized study. Am J Clin Nutr. 2014 Sep;100(3):813-20. doi: 10.3945/ajcn.113.081505. Epub 2014 Jul 23. PMID 25057155